CLINICAL TRIAL: NCT04887077
Title: Digital Intervention Promoting Physical Activity Among Obese People Randomized Controlled Trial: Assessing the Effects of a Digital Intervention to Promote Physical Activity in Patients With Obesity and/or Type 2 Diabetes Mellitus
Brief Title: Digital Intervention Promoting Physical Activity Among Obese People (DIPPAO)
Acronym: DIPPAO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: SENS laboratory, Univ. Grenoble Alpes (Unknown); INRAE, UNH, CRNH Auvergne, Clermont Auvergne University (Unknown); Kiplin (Unknown); I-SITE Clermont Auvergne Project 20-25 (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RBHP 2020 DUCLOS 2; 2020-A03091-38 (Other: ANSM)
Record Dates: First submitted 2021-05-03; First posted 2021-05-14 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Obesity; Diabete Type 2
Keywords: eHealth; Physical activity; Gamification; Mobile app; Behavior change; Cost-utility; Weight stigma
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Motor Activity; Weight Prejudice

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, controlled with two parallel arms.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Research assistants collecting data will be blinded to the treatment allocation. Double blinding is nevertheless not possible in such interventions because allocation concealment is impossible for participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kiplin intervention (Experimental): Kiplin intervention composed of the access to a mobile app and to telecoaching sessions. The number of teleocaching sessions per week will decrease over 3 months.
  Interventions: Device: Kiplin
- face-to-face supervised PA (usual care at the University Hospital of Clermont-Ferrand, France) (Active Comparator): three-month program of face-to-face adapted physical activity, three sessions a week, for a total of 36 sessions.
  Interventions: Behavioral: face-to-face

INTERVENTIONS:
Device: Kiplin — The Kiplin intervention will be composed of four components within a smartphone application: a) a gamification of Physical Activity through multiple games called "animations", b) a remote adapted physical activity program with telecoaching sessions, c) an interface for exchange and conversation and, d) an activity monitoring tool.
  Arms: Kiplin intervention
Behavioral: face-to-face — three-month program of face-to-face adapted physical activity, three sessions a week, for a total of 36 sessions.
  Arms: face-to-face supervised PA (usual care at the University Hospital of Clermont-Ferrand, France)

SUMMARY:
Overweight and obesity are today considered among the most important health risks facing humanity with more than one in two adults overweight or obese in western countries. In addition, Type 2 diabetes mellitus (T2DM) is a common comorbidity associated with overweight and obesity and counts for 5% of the French population under 65 years of age and 15% in people over 65 years old. Despite the accumulation of scientific evidence supporting the benefits of physical activity, obese and diabetic people remain insufficiently active and current programs struggle to engage and sustain physical activity of patients over long periods of time. It is therefore urgent to develop interventions that can effectively change individuals' behavior. In this context, "e-health" interventions and gamification appear to be a particularly promising avenue to improve physical activity and reduce attrition rates of current programs.

This clinical trial aim to test the effectiveness of a digital intervention based on gamification and teamwork in comparison to a supervised physical activity program. The investigators hypothesized that the intervention will be efficient by the development of a self-determined motivation through the process of gamification on the one hand. On the other hand, through the in-group collaboration with other people who share the same stigmatized criteria that will help participants to overcome weight stigmas, acting generally as physical activity barriers.

DETAILED DESCRIPTION:
This trial is a randomized, two-arm intervention design that will examine the efficacy of a digital group-based intervention based on gamification and teamwork among obese and T2DM patients. The experimental arm will be compared to an active control group representing the traditional care program (supervised physical activity).

The digital intervention is composed of four components within a smartphone application: a) a gamification of PA, b) a remote adapted physical activity program with telecoaching sessions, c) an interface for exchange and conversation and, d) an activity monitoring tool. Accelerometer data, self-reported PA, body composition, and physical capacities will be assessed before, at the end of the intervention and then at the issue of a 6-month follow up. To advance our understanding of complex interventions like gamified and group-based ones, this study will explore several psychological mediators relative to motivation, enjoyment, in-group identification, or perceived weight stigma. Finally, to assess a potential superior efficiency compared to the current treatment (face-to-face supervised PA), this study will include a cost-utility analysis between the two conditions.

ELIGIBILITY:
Inclusion Criteria:

* Subject affected for obesity (BMI ≥30 kg/m² and <45 kg/m²) and/or T2DM.
* Subject treated at the University Hospital of Clermont-Ferrand.
* The participants must have an iOS (at least iOS8 version) or Android (at least version 5) smartphone.
* Subjects must also be able to provide informed consent to participate in the research and be covered by health social security.
* Subjects must be native to any physical activity intervention.
* Sufficient proficiency of French will be required to ensure the understanding of the questionnaires.

Exclusion Criteria:

* Medical or surgical history judged by the investigator to be incompatible with the study.
* Subject with an unstable psychiatric condition.
* Pregnant or breastfeeding women.
* Heavy alcohol consumption (> 2 to 3 drinks per day depending on gender) or drug addiction.
* Disability or contraindication to PA.
* Subject with cardiorespiratory and/or osteoarticular disorders that limit their ability to perform physical tests or moderate PA for 30 minutes.
* Subject with progressive cardiovascular or neoplastic disease.
* Subject who has presented a major infection in the 3 months prior to inclusion.
* Subject with a known neuro-muscular pathology (i.e., myopathy, myasthenia, rhabdomyolysis, paraplegia, hemiplegia).
* Subject with chronic or acute inflammatory pathology within 3 months prior to inclusion.
* Subject diagnosed and/or treated for schizophrenia, bipolar disorder, major depression.
* Subject deprived of their liberty by judicial or administrative decision.
* Subject refusing to sign the written consent to participate.
* Subject participating in another study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
Change in daily physical activity from baseline to 3 months | Month 3
  The primary outcome will be the change of daily physical activity measured as the daily step count assessed via the Garmin Vivofit 3 (Garmin International Inc., Olathe, KS, USA)

SECONDARY OUTCOMES:
Change in body composition (BMI) from baseline to 9 months | Month 9
  in kg/m2
Change in body composition from baseline to 9 months | Month 9
  evaluated by bioelectrical impedance analysis
Change in daily physical activity from baseline to 9 months | Month 9
  measured as the daily step count assessed via the Garmin Vivofit 3 (Garmin International Inc., Olathe, KS, USA)
Change in physical activity level from baseline to 9 months | Month 9
  total physical activity (minutes/day) measured using the Garmin Vivofit 3 (Garmin International Inc., Olathe, KS, USA)
Change in moderate-to-vigorous physical activity (MVPA) from baseline to 9 months | Month 9
  measured using a tri-axial accelerometer (ActiGraph GT3x; ActiGraph LLC, Pensacola, FL, USA).
Change in light physical activity (LPA) from baseline to 9 months | Month 9
  measured using a tri-axial accelerometer (ActiGraph GT3x; ActiGraph LLC, Pensacola, FL, USA).
Change in sedentary time from baseline to 9 months | Month 9
  measured using a tri-axial accelerometer (ActiGraph GT3x; ActiGraph LLC, Pensacola, FL, USA).
Change in self-reported physical activity from baseline to 9 months | Month 9
  measured using the RPAQ
Change in six minute walking distance from baseline to 9 months | Month 9
  measured via the 6-minute walking test
Change in muscular strength of the upper limbs from baseline to 9 months | Month 9
  measured via handgrip measurements
Change in muscular strength of the lower limbs from baseline to 9 months | Month 9
  measured via isokinetic dynamometer
Programme adherence | Month 3
  number of APA sessions attended. Application engagement and utilization for the experimental group only
Change in quality of life from baseline to 9 months | Month 9
  measured via the EQ-5D
Cost-utility analysis | Month 9
  measured using incremental cost-effectiveness ratio between the average difference in cost and the average difference in effectiveness (QALY) observed between the two arms
Perceived enjoyment of physical activity at the end of the intervention | Month 3
  measured using the Physical Activity Enjoyment Scale (PACES)
Social identification at the end of the intervention | Month 3
  measured via the In-group identification questionnaire
Psychological needs satisfaction at the end of the intervention | Month 3
  measured via the Psychological Need Satisfaction in Exercise Scale (PNSES)
Change in motivation toward physical activity from baseline to 9 months | Month 9
  Autonomous and controlled motivation toward physical activity via the EMAPS.
Change in weight stigma concerns from baseline to 9 months | Month 9
  measured using the scale developed by Hunger and Major
Change in perceived daily discrimination from baseline to 9 months | Month 9
  measured via the everyday discrimination scale
Change in weight bias internalisation from baseline to 9 months | Month 9
  measured via the Modified Weight Bias Internalization Scale (WBIS-M)

OTHER OUTCOMES:
Perceived vulnerability toward COVID-19 | Month 9
  measured using the perceived vulnerability questionnaire
Perceived digitalization | Month 9
  measured using a single item
Perceived exertion during the APA sessions | Month 3
  measured via the Borg scale

CONTACTS AND LOCATIONS:
Overall Officials: Martine Duclos, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: Yes
We will share de-identified data associated with the collected samples by depositing these data at the Open Science Framework (OSF) repository. The storage will be in Germany (Frankfurt). Data will include demographic, anthropometric, and physical measurements along with data from questionnaires and intervention adherence. We agree that we will identify where the data will be available and how to access the data in any publications and presentations that we author about these data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available via a public OSF project that will be accessible by everyone. We agree to deposit outcome data into the OSF repository as soon as possible but no later than within two years after the completion of the trial or upon acceptance of the data for publication, or public disclosure of a submitted patent application, whichever is earlier.

REFERENCES:
- [Derived] Mazeas A, Chalabaev A, Blond M, Pereira B, Duclos M. Digital intervention promoting physical activity among obese people (DIPPAO) randomised controlled trial: study protocol. BMJ Open. 2022 Jun 16;12(6):e058015. doi: 10.1136/bmjopen-2021-058015. PMID 35710254